CLINICAL TRIAL: NCT04064788
Title: The Effect of the Modified Constraint-Induced Movement Therapy Administered on Consecutive or Intermittent Days on Upper Extremity Function in Individuals With Hemiparetic Cerebral Palsy
Brief Title: Modified Constraint-Induced Movement Therapy in Children With Hemiparetic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Sezen Tezcan, Principal Investigator, Abant Izzet Baysal University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-ST-01
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Spastic Hemiplegic Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Consecutive mCIMT group (Experimental): 6 hours / day, 10 consecutive days, 60 hours mKZHT + 2 days 45 minutes / day traditional physiotherapy
  Interventions: Other: Consecutive Modified Constraint-Induced Movement Therapy
- Intermittent mCIMT group (Experimental): 6 hours / day 2 days a week 5 weeks, a total of 60 hours mKZHT + 2 days 45 min / day traditional physiotherapy
  Interventions: Other: Intermittent Modified Constraint-Induced Movement Therapy
- Traditional physiotherapy control group (Active Comparator): 45 min / day, 2 days a week traditional physiotherapy
  Interventions: Other: Traditional physiotherapy

INTERVENTIONS:
Other: Consecutive Modified Constraint-Induced Movement Therapy — Consecutive mCIMT group received 6 hours per day mCIMT sessions for consecutive 10 days. Accompanied by a physiotherapist in 1 hour of the 6-hour restriction period, the family was guided within the remaining period and the activities were adapted to daily life.
  Arms: Consecutive mCIMT group
Other: Traditional physiotherapy — Traditional physiotherapy within a specific program
  Arms: Traditional physiotherapy control group
Other: Intermittent Modified Constraint-Induced Movement Therapy — Intermittent mCIMT group received mCIMT session 6 hours per day for 10 days, spread over 5 weeks (two days per week). Accompanied by a physiotherapist in 1 hour of the 6-hour restriction period, the family was guided within the remaining period and the activities were adapted to daily life.
  Arms: Intermittent mCIMT group

SUMMARY:
Cerebral palsy (CP) is defined as a non-progressive lesion of the developing foetal or infant brain and causes variety of motor, sensory and cognitive impairments. Hemiplegic CP is the most common type of CP in term infants, involving one half of the body. In these individuals, muscle tone is reduced, and there is an inability to perform quality upper extremity movements due to increased muscle tone, increased reflexes, weakness in antagonist muscles. Due to spasticity upper extremity is present in shoulder adduction and internal rotation, elbow flexion and pronation, wrist and fingers flexed and thumb in palm position. Spontaneous movements of the upper extremity are decreased and abnormal. These individuals have a reduced upper extremity function ranging from mild incompetence to almost no use of the hand.

Constraint-Induced Movement Therapy (CIMT) is designed to improve the function of the most affected limb by restricting the use of the less affected limb in individuals with unilateral upper extremity involvement and implementing an intensive motor learning-based training program. In pediatric subjects, modified CIMT (mCIMT), which is called a 'child-friendly technique', has been applied, which shows some differences from the form of CIMT in adults. In mCIMT, the restriction time was reduced, activities with the child were performed within a play frame, in the environment in which the child was accustomed, and restriction methods such as gloves, splint, sling were used. In the literature CIMT has been used mainly in children with hemiplegic CP in the pediatric population. However, there are many studies in the literature evaluating the efficacy of mCIMT in individuals with hemiplegic CP and showing beneficial effects on upper extremity speed and skills, and the duration of application restriction varies considerably.

The aim of the investigator's study was to determine the effect of consecutive or intermittent implementation of mCIMT on upper extremity function in children with hemiplegic CP. Thus, it will be determined whether the modification of the duration of administration in the pediatric population varies in treatment results.

DETAILED DESCRIPTION:
33 children with spastic hemiplegia age between 5-18 years will participate study. Children's gross motor skills classified with Gross Motor Classification Sysytem (GMFCS) and hand abilities classified with Manual Ability Classification System (MACS). The children divided into 3 groups, consecutive mCIMT group, intermittent mCIMT group, and traditional physiotherapy control group. The consecutive mCIMT group received mCIMT treatment for 10 consecutive days in addition to the conventional physiotherapy sessions. A sling used to restrict the noninvolved upper extremity. The unaffected upper extremities of the children restricted for 6 hours and activities performed by using shaping techniques under the guidance of same therapist. Within the remaining period, the family implemented the activities with his/her child that are determined by the therapist using the motor learning principles, appropriate to the age of the child and that he / she likes to do. The assessments performed for all three groups before, 10 days after and 5 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of hemiplegic CP
* 5-18 years of age
* MACS level I, II or III
* GMFCS level I
* To have sufficient communication skills
* To be able to extend the wrist at least 20 degrees
* Lack of severe spasticity to prevent grasping and dropping objects
* Surgery or application of Botulinum toxin within the last 6 months
* The family's acceptance of the child's participation in the study
* The child volunteers to participate in the study

Exclusion Criteria:

* Visual and hearing impairment
* Family refuses to participate in the study
* There is a walking and balance problem that may cause a fall risk during the use of a sling
* Behavioral problems at the level to reject the practices to be performed within the study

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Children's Hand-Use Experience Questionnaire (CHEQ) | Change from Baseline at 10 days and at 5 weeks
  Assessing children's experience of using the affected hand in activities of daily living where usually two hands are needed. There are 29 items at questionnaire. When respondents answered the questionnaire, they were first asked whether the activity included in the questionnaire was conducted independently. If the activities can be done independently, it is questioned whether one or two hands are used during the activities. If two hands are used, answers and scores to the following 3 sub-questions are sought: hand use, time use in comparison to peers, experience of feeling bothered while doing the activity. A higher score indicates a better level of independence.
Jebsen-Taylor Hand Function Test | Change from Baseline at 10 days and at 5 weeks
  This is an objective test to evaluate hand function for a person's activities of daily living. Test consist of 7 subtests includes writing, card turning, manipulate small common objects, simulated feeding, stacking checkers, moving large light objects and moving large heavy objects. We will use 6 subtests except writing in our study.

SECONDARY OUTCOMES:
Gross Motor Classification System (GMFCS) | At Baseline
  This is a classification system for children with chronic disability and based on the movements initiated by the child him/herself such as sitting, moving and acting. GMFCS classifies gross motor functions of children with CP in five levels.
Manual Ability Classification System (MACS) | At Baseline
  MACS is a five-level classification system that analyzes the children with CP use their hands while carrying objects in their daily activities.
Pediatric Balance Scale (PBS) | At Baseline
  Assesses children's balance and consist of 14 items. Each item is scored between 0 and 4 points. Low score refers to the poor balance and the high score refers to the good balance.
Modified Tardieu Scale (MTS) | Change from Baseline at 10 days and at 5 weeks
  The scale was developed to evaluate spasticity. This scale reveals the rate-dependent nature of spasticity (27). Muscle reaction quality (X) and muscle reaction angle (Y) are determined with MTS. When measuring the muscle reaction angle, the goniometer is used to measure the position of the muscle with minimum stretching. If quality of muscle reaction score was 2 or higher, the joint angle in which the muscle responds with difficulty will be measured goniometer. The scales scores range from 0 to 5. 0= no resistance to passive movement. 1= slight resistance throughout the course of the passive movement. 2= there's a clear catching at a precise angle, which makes passive movement difficult, followed by a release. 3= fatigable clonus (Less than 10 seconds). 4= infatigable clonus (More than 10 seconds). 5= the joint cannot be moved. Evaluations are made in thre
ABILHAND-Kids Questionnaire | Change from Baseline at 10 days and at 5 weeks
  Evaluates manual ability in children with cerebral palsy. Questionnaire consist of 21 bimanual items. Each item graded three levels (0=impossible, 1= difficult, 2= easy) and lower scores indicate lower ability of the hand or upper extremity.
Surface electromyography (sEMG) | Change from Baseline at 10 days and at 5 weeks
  sEMG evaluates electrical activity of muscle groups. It is a non-invasive method used to evaluate muscle activation. Delsys Trigno Wireless System device will be used for measurements. Measurements using silver-silver chloride (Ag-AgCl) disposable adhesive electrodes will be performed in accordance with the criteria of SENIAM (surface EMG for non-invasive assessment of muscle) and literature.
Pediatric Evaluation of Disability Inventory (PEDI) | Change from Baseline at 10 days and at 5 weeks
  PEDI evaluates disability, activity and participation in pediatric population. It consist of 197 items and each item scored in the way 0: can not do, 1: can do.

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Çankaya, Study Director — Abant Izzet Baysal University; Sezen Tezcan, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

REFERENCES:
- [Background] Taub E, Ramey SL, DeLuca S, Echols K. Efficacy of constraint-induced movement therapy for children with cerebral palsy with asymmetric motor impairment. Pediatrics. 2004 Feb;113(2):305-12. doi: 10.1542/peds.113.2.305. PMID 14754942
- [Background] Brady K, Garcia T. Constraint-induced movement therapy (CIMT): pediatric applications. Dev Disabil Res Rev. 2009;15(2):102-11. doi: 10.1002/ddrr.59. PMID 19489088
- [Background] Hoare BJ, Wasiak J, Imms C, Carey L. Constraint-induced movement therapy in the treatment of the upper limb in children with hemiplegic cerebral palsy. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD004149. doi: 10.1002/14651858.CD004149.pub2. PMID 17443542
- [Background] Stearns GE, Burtner P, Keenan KM, Qualls C, Phillips J. Effects of constraint-induced movement therapy on hand skills and muscle recruitment of children with spastic hemiplegic cerebral palsy. NeuroRehabilitation. 2009;24(2):95-108. doi: 10.3233/NRE-2009-0459. PMID 19339749